CLINICAL TRIAL: NCT04163900
Title: A Phase III Open-Label, Multi-Centre, Randomized Study Comparing NUC-1031 Plus Cisplatin to Gemcitabine Plus Cisplatin in Patients With Previously Untreated Locally Advanced or Metastatic Biliary Tract Cancer
Brief Title: Comparing NUC-1031 Plus Cisplatin to Gemcitabine Plus Cisplatin in Patients With Advanced Biliary Tract Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A pre-planned futility analysis concluded that NUC-1031 plus cisplatin was unlikely to achieve its primary objective of improving overall survival. Based on the IDMC's recommendation, NuCana has closed the study.
Sponsor: NuCana plc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NuTide:121; 2019-001025-28 (EudraCT Number)
Record Dates: First submitted 2019-11-01; First posted 2019-11-15 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Biliary Tract Cancer
Keywords: Adenocarcinoma; Ampullary; Antineoplastic Agents; Biliary Tract Cancer; Chemotherapy; Cholangiocarcinoma; Cisplatin; Digestive System Neoplasms; Distal Bile Duct; Extrahepatic; First-line Chemotherapy; Gallbladder; Gastrointestinal; Gemcitabine; Hepatobiliary; Intrahepatic; Locally advanced; Metastatic; Neoplasm; NUC-1031; ProTides; Untreated
MeSH Terms: conditions — Biliary Tract Neoplasms; Adenocarcinoma; Cholangiocarcinoma; Digestive System Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — NUC-1031; Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: 1:1 randomization model to either Arm A or Arm B
Who Masked: Outcomes Assessor
Masking Description: Imaging scans will be assessed by blinded independent review according to RECIST v1.1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A - NUC-1031 and cisplatin (Experimental): 725 mg/m^2 NUC-1031 administered in combination with 25 mg/m^2 cisplatin on Days 1 and 8 of a 21-day cycle
  Interventions: Drug: NUC-1031; Drug: Cisplatin
- B - gemcitabine and cisplatin (Active Comparator): 1000 mg/m^2 gemcitabine administered in combination with 25 mg/m^2 cisplatin on Days 1 and 8 of a 21-day cycle
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: NUC-1031 — IV infusion in 500 mL of 0.9% sterile saline for injection given over 30 minutes
  Other Names: fosgemcitabine palabenamide
  Arms: A - NUC-1031 and cisplatin
Drug: Gemcitabine — IV infusion in 250 mL of 0.9% sterile saline for injection given in accordance with the package insert
  Other Names: Difluorodeoxycytidine; Gemzar
  Arms: B - gemcitabine and cisplatin
Drug: Cisplatin — IV in accordance with local institutional practice for biliary tract cancer, including the use of an appropriate hydration protocol
  Other Names: CDDP

SUMMARY:
NuTide:121 compares NUC-1031 with gemcitabine, both in combination with cisplatin, in patients with previously untreated advanced biliary tract cancer.

The primary hypotheses are:

* The combination of NUC-1031 plus cisplatin prolongs overall survival compared to the gemcitabine plus cisplatin standard of care
* The combination of NUC-1031 plus cisplatin increases overall response rate compared to the gemcitabine plus cisplatin standard of care

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and authorization to use and disclose health information.
2. Ability to comprehend and willingness to comply with the requirements of this protocol, including the QoL questionnaires.
3. Female or male patients aged ≥18 years.
4. Histologically- or cytologically-confirmed adenocarcinoma of the biliary tract (including gallbladder, intra and extra-hepatic biliary ducts and ampullary cancers) that is locally advanced, unresectable or metastatic (AJCC edition 8, 2018). Patients with measurable (as per RECIST v1.1 criteria) or non-measurable disease are permitted.
5. Life expectancy ≥16 weeks.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Adequate biliary drainage with no evidence of ongoing infection. If applicable, treatable and clinically-relevant biliary duct obstruction has been relieved by internal endoscopic drainage/stenting at least 2 weeks previously or by palliative bypass surgery or percutaneous drainage prior to study treatment, and the patient has no active or suspected uncontrolled infection. Patients fitted with a biliary stent should be clinically stable and free of signs of infection for ≥2 weeks prior to study treatment. Patients with improving biliary function who meet all other inclusion criteria may be re-tested during the screening window.
8. Adequate bone marrow, hepatic, and renal function, as evidenced by:

   * Absolute neutrophil count (ANC) ≥1,500/μL without colony-stimulating factor support
   * Platelet count ≥100,000/μL
   * Haemoglobin ≥9 g/dL without need for haematopoietic growth factor or transfusion support in prior 2 weeks
   * Total bilirubin <2 × upper limit of normal (ULN); does not apply to patients with Gilbert's syndrome. Consistent with inclusion criterion 7, patients whose whole bilirubin and biliary function is recovering may be re-tested during the screening period.
   * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) <5 × ULN
   * Creatinine clearance ≥45 mL/min actual or calculated by the Cockcroft-Gault method
   * International normalized ratio (INR) <1.5 and activated partial thromboplastin time (aPTT) <1.5 × ULN; does not apply to patients on an anti-coagulant with stable dose 28 days prior to first dose.
9. QTc interval <450 msec (males) or <470 msec (females), in the absence of bundle branch block. In the presence of bundle branch block with consequent QTc prolongation, patients may be enrolled based on a careful risk-benefit assessment.
10. Human Immunodeficiency Virus-infected patients who are healthy and have a low risk of Acquired Immunodeficiency Syndrome-related outcomes may be included in this study.
11. Female patients of child-bearing potential (i.e., all women except those who are post-menopausal for ≥1 year or who have a history of hysterectomy or surgical sterilization) must have a negative pregnancy test within 3 days prior to the first study drug administration. All patients of child-bearing potential must agree to practice true abstinence or to use two highly effective forms of contraception, one of which must be a barrier method of contraception, from the time of screening until 6 months after the last dose of study medication.
12. Male patients with a female partner must either have had a successful vasectomy or they and their female partner meet the criteria above (not of childbearing potential or practicing highly effective contraceptive methods).

Exclusion Criteria:

1. Combined or mixed hepatocellular/cholangiocarcinoma.
2. Prior systemic therapy for advanced or metastatic biliary tract cancer. However, prior chemotherapy in the adjuvant setting or low-dose chemotherapy given in conjunction with radiotherapy in the adjuvant setting and completed at least 6 months prior to enrolment is permitted. The following prior interventions are allowed provided the patient has fully recovered:

   * Surgery: non-curative resection with macroscopic residual disease or palliative bypass surgery. Patients who have previously undergone curative surgery must now have evidence of non-resectable disease requiring systemic chemotherapy.
   * Radiotherapy: prior radiotherapy (with or without radio-sensitizing low-dose chemotherapy) for localized disease and there is now clear evidence of disease progression requiring systemic chemotherapy.
   * Photodynamic therapy: prior photodynamic therapy for localized disease with no evidence of metastatic disease or for localized disease to relieve biliary obstruction in the presence of metastatic disease provided there is now clear evidence of disease progression requiring systemic chemotherapy.
   * Palliative radiotherapy: palliative radiotherapy provided that all adverse events have resolved and the patient has measurable disease outside the field of radiation.
3. Prior treatment with or known hypersensitivity to NUC-1031, gemcitabine, cisplatin or other platinum-based agents or history of allergic reactions attributed to any parenteral excipients (e.g. dimethylacetamide [DMA], Cremophor EL, Polysorbate 80, Solutol HS 15).
4. Symptomatic central nervous system or leptomeningeal metastases.
5. History of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, surgically excised or potentially curatively treated ductal carcinoma in situ of the breast, or low grade prostate cancer or patients after prostatectomy not requiring treatment. Patients with previous invasive cancers are eligible if treatment was completed more than 3 years prior to initiating the current study treatment, and the patient has had no evidence of recurrence since then.
6. Concurrent serious (as deemed by the Investigator) medical conditions, including, but not limited to, New York Heart Association class III or IV congestive heart failure, history of congenital prolonged QT syndrome, uncontrolled infection, active hepatitis B or C, or other co-morbid conditions that in the opinion of the Investigator would impair study participation or cooperation.
7. Congenital or acquired immunodeficiency (e.g., serious active infection with HIV). As per inclusion criterion 10, patients with HIV who are healthy and have a low risk of AIDS related outcomes are eligible.
8. Other acute or chronic medical, neurological, or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.
9. Prior exposure to another investigational agent within 28 days prior to randomization.
10. Major surgery within 28 days prior to randomization; patient must have completely recovered from any prior surgical or other procedures.
11. Pregnant or breastfeeding.
12. Residual toxicities from prior treatments or procedures which have not regressed to Grade ≤1 severity (CTCAE v5.0), except for alopecia or ≤ Grade 2 peripheral neuropathy.
13. Concomitant use of drugs at doses known to cause clinically relevant prolongation of QT/QTc interval.
14. Administration of a live vaccination within 28 days prior to randomization.
15. Ongoing or recent (≤6 months) hepatorenal syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 773 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knox, MD, Principal Investigator — Professor of Medicine, University of Toronto
Locations (125):
- United States (29):
  - Arizona Oncology Associates , PC - HOPE, Tucson, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Rocky Mountain Cancer Centers, LLP- Aurora, Aurora, Colorado
  - Baptist Health Medical Group Oncology, LLC, Miami, Florida
  - Orlando Health, Inc., Orlando, Florida
  - IACT Health, Columbus, Georgia
  - Affiliated Oncologists LLC, Chicago Ridge, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Medical Group, Detroit, Michigan
  - Minnesota Oncology Hemtology, Minneapolis, Minnesota
  - Regents of the University of Minnesota, Minneapolis, Minnesota
  - University of Rochester Medical Center - Strong Memorial Hospital, Rochester, New York
  - The Research Foundation for The State University of New York, Stony Brook, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, Pennsylvania
  - Prisma Health Upstate, Greenville, South Carolina
  - Texas Oncology, P.A. - Austin, Austin, Texas
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Texas Oncology, P.A. - Tyler, Tyler, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Northwest Cancer Specialists, P.C.-Vancouver, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Australia (9):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Newcastle Private Hospital, Newcastle, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Townsville Cancer Centre, Townsville, Queensland
  - Warringal Medical Centre, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHUM Centre de Recherche, Montreal, Quebec
  - SMBD Jewish General Hospital, Montreal, Quebec
- Czechia (5):
  - Fakultní nemocnice Brno, Brno
  - Fakultní nemocnice Hradec Králové, Hradec Králové
  - Fakultní nemocnice Olomouc, Olomouc
  - Thomayerova nemocnice, Prague
  - Nemocnice Na Homolce, Prague
- France (5):
  - Centre Georges François Leclerc, Dijon
  - CHU de Grenoble - Hôpital Nord, Grenoble
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Hôpital Cochin, Paris
  - ICO - Site René Gauducheau, Saint-Herblain
- Germany (5):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Vivantes Klinikum Neukoelln, Berlin
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Tuebingen, Tübingen
- Hungary (6):
  - Semmelweis Egyetem, Budapest
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem, Debrecen
  - Borsod-Abauj-Zemplen Megyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Italy (6):
  - Ospedale Policlinico San Martino, Genova
  - IEO Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Centro Ricerche Cliniche di Verona S.r.l, Verona
- Russia (7):
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow
  - FSBSI Russian Oncological Scientific Center n.a. N.N. Blokhin, Moscow
  - "VitaMed" LLC, Moscow
  - State Budget Institution of Healthcare "Leningrad Regional Clinical Oncology Dispensary", Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - SPb SBIH "City Clinical Oncological Dispensary", Saint Petersburg
  - Medicinskiy gorod, Tyumen
- South Korea (10):
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Dong-A University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
- Spain (9):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario HM Madrid Sanchinarro, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (5):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - MacKay Medical Foundation The Presbyterian Church in Taiwan MacKay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (7):
  - Acibadem Adana Hospital, Adana
  - Baskent University Adana Application and Research Center, Adana
  - Akdeniz University Medical Faculty, Antalya
  - Trakya University Medical Faculty, Edirne
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Dr. Abdurrahman Yurtaslan Oncology Teaching and Research Hospital, Malatya
  - Inonu University Medical Facility, Malatya
- Ukraine (8):
  - CI Chernivtsi RC Oncological Dispensary, Chernivtsi
  - Communal Non-profit Enterprise Regional Center of Oncology, Kharkiv NMU, Kharkiv
  - CI of Healthcare Regional Clinical Specialized Dispensary of the Radiation Protection, Kharkiv
  - Kyiv City Clinical Oncological Center, Kyiv
  - SI "Shalimov's National Institute of Surgery and Transplantation" of NAMSU, Kyiv
  - Treatment-Prevention Institution Volyn Regional Oncological Dispensary, Lutsk
  - Communal Institution Odesa Regional Clinical Hospital, Odesa
  - RCI Sumy Regional Clinical Oncological Dispensary, Sumy
- United Kingdom (6):
  - Guy's Hospital, London, Greater London
  - The Christie, Manchester, Greater Manchester
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knox JJ, McNamara MG, Bazin IS, Oh DY, Zubkov O, Breder V, Bai LY, Christie A, Goyal L, Cosgrove DP, Springfeld C, Sjoquist KM, Park JO, Verdaguer H, Braconi C, Ross PJ, De Gramont A, Shroff RT, Zalcberg JR, Palmer DH, Smith JR, Oelmann E, Bruce T, Valle JW. A phase III randomized study of first-line NUC-1031/cisplatin vs. gemcitabine/cisplatin in advanced biliary tract cancer. J Hepatol. 2025 Aug;83(2):358-366. doi: 10.1016/j.jhep.2025.01.040. Epub 2025 Feb 18. PMID 39978598
- [Derived] McNamara MG, Goyal L, Doherty M, Springfeld C, Cosgrove D, Sjoquist KM, Park JO, Verdaguer H, Braconi C, Ross PJ, Gramont A, Zalcberg JR, Palmer DH, Valle JW, Knox JJ. NUC-1031/cisplatin versus gemcitabine/cisplatin in untreated locally advanced/metastatic biliary tract cancer (NuTide:121). Future Oncol. 2020 Jun;16(16):1069-1081. doi: 10.2217/fon-2020-0247. Epub 2020 May 6. PMID 32374623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 773 patients were recruited between Dec 2019 and March 2022.
Period: Overall Study
Arm/Group | A - NUC-1031 and Cisplatin | B - Gemcitabine and Cisplatin
Started | 388 | 385
Received Study Treatment (Safety Population) | 383 | 378
Completed | 0 | 0
Not Completed | 388 | 385
Not completed — Radiological disease progression | 112 | 127
Not completed — Study closure | 98 | 133
Not completed — Adverse Event | 78 | 32
Not completed — Withdrawal by Subject | 37 | 34
Not completed — Death | 29 | 16
Not completed — Physician Decision | 17 | 25
Not completed — Clinical disease progression | 14 | 13
Not completed — Protocol Violation | 3 | 4
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | A - NUC-1031 and Cisplatin | B - Gemcitabine and Cisplatin | Total
Number analyzed (Participants) | 388 | 385 | 773
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 185 | 186 | 371
  >=65 years | 203 | 199 | 402
Age, Continuous [Median (Full Range); unit: years] | 65.0 [31 to 87] | 65.0 [20 to 86] | 65.0 [20 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 188 | 362
  Male | 214 | 197 | 411
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 31 | 52
  Not Hispanic or Latino | 359 | 337 | 696
  Unknown or Not Reported | 8 | 17 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 76 | 77 | 153
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 5 | 8
  White | 285 | 274 | 559
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 23 | 28 | 51
Primary tumour location [Count of Participants; unit: Participants]
  Gallbladder | 80 | 80 | 160
  Intra-hepatic | 209 | 207 | 416
  Extra-hepatic | 80 | 80 | 160
  Ampullary | 19 | 18 | 37
Extent of disease [Count of Participants; unit: Participants]
  Locally advanced | 56 | 65 | 121
  Metastatic | 330 | 320 | 650
  Unknown | 2 | 0 | 2
Measurable disease [Count of Participants; unit: Participants] — Patients with measurable disease as determined by RECIST v1.1 criteria:
  Tumour lesions must be accurately measured in at least one dimension (longest diameter in the plane of measurement to be recorded) with a minimum size of:
  * 10 mm by CT or MRI scan (CT/MRI scan slice thickness/interval no greater than 5 mm)
  * 10-mm caliper measurement by clinical examination
  To be considered pathologically enlarged and measurable, a lymph node must be ≥15 mm in the short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm).
  Participants
    Yes | 367 | 366 | 733
    No | 21 | 19 | 40
ECOG performance status [Count of Participants; unit: Participants] — The ECOG score describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). The score runs from 0 to 5, with 0 denoting perfect health and 5 death. Patients with scores of 0 or 1 were eligible for this study:
  0 - Asymptomatic. Fully active, able to carry on all predisease activities without restriction
  1 - Symptomatic but completely ambulatory. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Participants
    0 | 205 | 186 | 391
    1 | 178 | 192 | 370
    Unknown | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Percentage of patients achieving a confirmed complete response (CR) or partial response (PR) to treatment as assessed by blinded independent review according to RECIST v1.1 criteria. ORR = patients with CR + patients with PR, where" CR = disappearance of all target lesions PR = at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters This outcome was assessed in the population of patients with measurable disease at baseline who were also randomized ≥28 weeks before the data cut-off (ITTMD28). Patients were to receive a confirmatory scan 28-42 days after response is first observed.
Time Frame: Evaluated at Screening (baseline) then every 9 weeks from treatment start (C1D1), or every 12 weeks if treatment is stopped with no evidence of progression, until disease progression or death from any cause up to the end of study, an average of 6 months.
Population: Intent-to-treat with measurable disease at baseline randomized ≥28 weeks before the data cut-off (ITTMD28)
Measure: Count of Participants; unit: Participants
Arm/Group | A - NUC-1031 and Cisplatin | B - Gemcitabine and Cisplatin
Number analyzed (Participants) | 284 | 275
Participants | 53 | 34

2. Primary Outcome: Overall Survival (OS)
Description: The median time, in months, from the date of randomization to the date of death from any cause. For patients who were alive at the time of a data cut-off or were permanently lost to follow up, duration of OS was censored at the date at which they were last known to be alive.
Time Frame: From the date of randomization until the date of death from any cause, assessed up to 12 months on average
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | A - NUC-1031 and Cisplatin | B - Gemcitabine and Cisplatin
Number analyzed (Participants) | 388 | 385
Months | 9.2 [8.3 to 10.4] | 12.6 [11.0 to 15.1]

ADVERSE EVENTS:
Time Frame: Each patient was assessed for serious and other (non-serious) adverse events from the date of consent until 30 days after the last dose of study treatment, an average of 6 months. Each patient was assessed for all-cause mortality from the date of randomization until the date of death from any cause, an average of 12 months
Description: All adverse events are reported for the Safety Population, which consisted of all patients in the ITT population who also received any study medication. This differs from all-cause mortality, which is reported for the ITT population.
Arm/Group | A - NUC-1031 and Cisplatin | B - Gemcitabine and Cisplatin
All-Cause Mortality (participants affected / at risk) | 188/388 | 135/385
Serious Adverse Events (participants affected / at risk) | 175/383 | 126/378
Other Adverse Events (participants affected / at risk) | 370/383 | 369/378
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A - NUC-1031 and Cisplatin (N=383) | B - Gemcitabine and Cisplatin (N=378)
Sepsis (Infections and infestations) | 12 | 12
pneumonia (Infections and infestations) | 5 | 5
Biliary sepsis (Infections and infestations) | 5 | 3
Biliary tract infection (Infections and infestations) | 3 | 5
COVID-19 (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 4 | 3
Bacteraemia (Infections and infestations) | 2 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 2
Pseudomonal sepsis (Infections and infestations) | 1 | 2
COVID-19 pneumonia (Infections and infestations) | 1 | 2
Device related infection (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 1 | 1
Liver abscess (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Neutropenic sepsis (Infections and infestations) | 0 | 2
Peritonitis (Infections and infestations) | 1 | 1
Spontaneous bacterial peritonitis (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bacillus bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Clostridium bacteraemia (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Device related bacteraemia (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1
Epiglottitis (Infections and infestations) | 1 | 0
Gallbladder abscess (Infections and infestations) | 0 | 1
Hepatitis B reactivation (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 0 | 1
Suspected COVID-19 (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 12 | 18
Asthenia (General disorders) | 2 | 3
Fatigue (General disorders) | 5 | 0
General physical health deterioration (General disorders) | 4 | 1
Oedema peripheral (General disorders) | 4 | 1
Death (unknown cause) (General disorders) | 2 | 2
Generalised oedema (General disorders) | 2 | 1
Gait disturbance (General disorders) | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Discomfort (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 9
Ascites (Gastrointestinal disorders) | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 3 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Subileus (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Jejunal ulcer (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 8 | 4
Biliary obstruction (Hepatobiliary disorders) | 5 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 4 | 2
Hepatic failure (Hepatobiliary disorders) | 5 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 2
Cholangitis acute (Hepatobiliary disorders) | 2 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 3 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 0
Jaundice (Hepatobiliary disorders) | 3 | 0
Gallbladder rupture (Hepatobiliary disorders) | 1 | 1
Liver injury (Hepatobiliary disorders) | 2 | 0
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0
Hepatic vein embolism (Hepatobiliary disorders) | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Portal vein embolism (Hepatobiliary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 5
Platelet count decreased (Investigations) | 4 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Cytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 7 | 2
Embolism (Vascular disorders) | 2 | 2
Embolism arterial (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 1 | 1
Arterial thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 2
Ischaemic stroke (Nervous system disorders) | 1 | 4
Hepatic encephalopathy (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Device occlusion (Product Issues) | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Personality change (Psychiatric disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A - NUC-1031 and Cisplatin (N=383) | B - Gemcitabine and Cisplatin (N=378)
Nausea (Gastrointestinal disorders) | 167 | 142
Alanine aminotransferase increased (Investigations) | 142 | 62
Fatigue (General disorders) | 139 | 114
Aspartate aminotransferase increased (Investigations) | 121 | 57
Constipation (Gastrointestinal disorders) | 105 | 102
Anaemia (Blood and lymphatic system disorders) | 99 | 183
Neutropenia (Blood and lymphatic system disorders) | 88 | 133
Vomiting (Gastrointestinal disorders) | 81 | 65
Thrombocytopenia (Blood and lymphatic system disorders) | 76 | 74
Platelet count decreased (Investigations) | 67 | 63
Blood bilirubin increased (Investigations) | 66 | 17
Asthenia (General disorders) | 64 | 63
Edema peripheral (General disorders) | 61 | 52
Hypomagnesemia (Metabolism and nutrition disorders) | 64 | 59
Decreased appetite (Metabolism and nutrition disorders) | 59 | 55
Abdominal pain (Gastrointestinal disorders) | 53 | 52
Neutrophil count decreased (Investigations) | 57 | 83
Pyrexia (General disorders) | 37 | 45
Diarrhea (Gastrointestinal disorders) | 48 | 56
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 27
Ascites (Gastrointestinal disorders) | 32 | 13
Hypoalbuminemia (Metabolism and nutrition disorders) | 39 | 22
Leukopenia (Blood and lymphatic system disorders) | 23 | 40
Abdominal pain upper (Gastrointestinal disorders) | 19 | 36
Dyspepsia (Gastrointestinal disorders) | 21 | 20
Abdominal distension (Gastrointestinal disorders) | 22 | 14
Blood alkaline phosphatase increased (Investigations) | 36 | 26
White blood cell count decreased (Investigations) | 25 | 33
Weight decreased (Metabolism and nutrition disorders) | 20 | 25
Blood creatinine increased (Metabolism and nutrition disorders) | 9 | 24
Hypokalaemia (Metabolism and nutrition disorders) | 27 | 21
Hyperglycemia (Metabolism and nutrition disorders) | 22 | 20
COVID-19 (Infections and infestations) | 20 | 17
Dizziness (Nervous system disorders) | 37 | 27
Headache (Nervous system disorders) | 30 | 29
Dysgeusia (Nervous system disorders) | 25 | 24
Neuropathy peripheral (Nervous system disorders) | 9 | 24
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 34 | 32
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 26
Hypertension (Vascular disorders) | 19 | 26
Deep vein thrombosis (Vascular disorders) | 18 | 13
Hyperbilirubinemia (Hepatobiliary disorders) | 31 | 8
Insomnia (Psychiatric disorders) | 19 | 32
Infusion related reaction (Injury, poisoning and procedural complications) | 19 | 2

LIMITATIONS AND CAVEATS:
At Interim Analysis 1, the futility boundary for OS was crossed and the study was closed on 02 Mar 2022. Following study closure, data from the 05 April 2022 final data cut-off (30 day follow-up post the last patient last visit) were analysed. In general, the analyses performed on this final database were those that were scheduled to take place at Interim Analysis 2. However, any p-values or CIs obtained are only viewed as descriptive as the study was stopped for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT04163900/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT04163900/SAP_001.pdf